CLINICAL TRIAL: NCT05489978
Title: Effectiveness of a Cervical Cancer Stigma Reduction Intervention Program on Cancer Stigma Score and Cervical Cancer Screening Uptake in Nepal- A Cluster Randomised Controlled Trial
Brief Title: Effectiveness of a Cervical Cancer Stigma Reduction Intervention Program on Cancer Stigma Score and Cervical Cancer Screening Uptake in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Priyanka Timsina, Student, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CC2022
Record Dates: First submitted 2022-05-24; First posted 2022-08-05 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Cervical Cancer; Stigma; Screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Randomization will allocate women to intervention and control arm in 1:1 ratio; with 6 wards in each group. The intervention arm will consist of 153 women who will receive "Cervical Cancer Stigma Reduction Intervention".
  Interventions: Behavioral: "Cervical Cancer Stigma Reduction Intervention"
- Control Arm (No Intervention): The control arm will consist of 153 women who would not be given any intervention.

INTERVENTIONS:
Behavioral: "Cervical Cancer Stigma Reduction Intervention" — Change in knowledge:
  Cervical cancer burden in Nepal, signs and symptoms, preventive measures available, lifestyle modifications, HPV vaccination, early diagnosis, screening, and treatment.
  Change in Stigma
  1. Para-social contact
     * Video of a person facing cervical cancer what symptoms she got, how she dealt with it, and how she overcame it.
     * Experiences of a cervical cancer survivor so that women personalize the information by relating it to their own life experiences by changing their attitude and behavior.
  2. Participatory learning techniques
     * Personal stories: Voluntary self-reflection of any stigma they perceive on cervical cancer or their community perceives cervical cancer.
     * Group Discussion: Discuss the drivers of stigma, facilitators of sigma, types of stigma prevalent in your community, and consequences of stigma.
  3. Myths vs facts: Negative attitudes, myths, and misconceptions about cervical cancer will be contraindicated by factual information.
  Arms: Intervention Arm

SUMMARY:
It is a cluster randomized control trial to assess the effectiveness of the cervical cancer stigma reduction intervention on cancer stigma score and cervical cancer screening uptake in Nepal

DETAILED DESCRIPTION:
Despite the presence of ample evidence, that stigma is one of the major reasons for low screening coverage, Nepal does not have a single stigma reduction intervention targeted among women to increase cervical cancer screening coverage. Therefore, we aim to assess the effectiveness of a stigma reduction education program on stigma score and cervical cancer screening uptake in Nepal. We will conduct a two-arm open-label cluster-interventional study in Budanilkhantha Municipality. A computer-based program will randomly allocate the 12 wards of Budanilkhantha Municipality with an allocation ratio 1:1; 6 wards in intervention group and 6 wards in control group. We will conduct a "stigma reduction education program" in the intervention group. After that we will follow up the participants for2 months to see the effectiveness of a stigma reduction education program on stigma score and cervical cancer screening uptake in Nepal. We will analyze data using STATA 14. We will use independent tests to find the mean difference between cervical cancer screening uptake and cervical cancer stigma score. The difference in mean among the two groups will actually be the difference due to intervention given. Findings from this study will help managers and stakeholders to formulate and improve strategies on screening programs and develop programs to reduce stigma on cervical cancer among women in Nepal.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30-60 years (the age range recommended for VIA screening in Nepal
* Married women
* Residents of Budanilkantha Municipality

Exclusion Criteria:

* Women who have already undergone screening within 5 years.
* Women with hearing or mental disorders
* Pregnant women
* Less than 6 weeks postpartum
* Mothers who had lived in the community for less than 6 months to perform seasonal work (e.g. in brick kilns) or visitors in the family.
* Women who are already diagnosed with cervical pre-cancer and cancer and have undergone hysterectomy.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study population will be women aged 30-60 years which is the recommended age group by National Guideline for Cervical Cancer Screening and Prevention in Nepal
Enrollment: 310 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Mean stigma score | Measured at baseline and endline (after 2 months gap from baseline)
  Change in mean stigma score using Cancer Stigma Scale at baseline and follow up

SECONDARY OUTCOMES:
Cervical cancer screening uptake | Measured within a month after endline
  Number of women attending cervical cancer screening program in intervention and control groups

CONTACTS AND LOCATIONS:
Locations (1):
- Budanilkantha Municipality, Kathmandu, Province-3, Nepal

IPD SHARING:
Plan to Share IPD: No